CLINICAL TRIAL: NCT06896526
Title: Comprehensive Outcomes Monitoring for Peri- and Postnatal Invasive Group B Strep Sequelae (COMPPASS) Registry
Acronym: COMPPASS
Status: Not yet recruiting | Type: Observational
Sponsor: Precia Group (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-2025-IG
Record Dates: First submitted 2025-03-03; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Invasive Group B Streptococcus Disease; Group B Streptococcus; Group B Streptococcal Infection; Group B Streptococcus (GBS) Disease; Group B Streptococcal Infection, Early-Onset; Group B Streptococcal Infection, Late-Onset
Keywords: Invasive Group B Streptococcus Disease; Invasive Group B Streptococcus Registry
MeSH Terms: conditions — Streptococcal Infections; Guillain-Barre Syndrome; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this registry is to collect and store important medical and non-health information on children from 0 to 18 years of age affected by early- (up to 24 hours after birth) and late-onset (up to 90 days after birth) invasive Group B Streptococcus (iGBS) and their families. Data collected from families of children affected by perinatal iGBS will support further research to understand the short- and long-term impact of iGBS disease on affected children and its impact on their families. Participants will be invited to complete obstetric and pregnancy-related questionnaires as well as validated neurodevelopmental surveys at various timepoints throughout their participation in the registry.

DETAILED DESCRIPTION:
BACKGROUND Group B Streptococcus (GBS) is a bacterial pathogen and the leading cause of severe neonatal infections and neonatal mortality, maternal morbidity, and adverse pregnancy outcomes globally. If not treated, Group B streptococcus (GBS) colonization during pregnancy can lead to invasive GBS disease (iGBS) in infants, including meningitis or sepsis, with a high mortality risk. Surviving infants have a higher risk of long-term neurodevelopmental impairment (NDI), especially with meningitis, though it is now understood that NDI after iGBS sepsis has been underestimated and is considered a current data gap. The purpose of this registry is to collect clinical and non-clinical data related to diagnosis and parent reported outcomes of their surviving infants related to long-term NDI.

SIGNIFICANCE Understanding the burden of NDI in this population may help identify opportunities for early screening and intervention for NDI, as interventions are likely to be more effective when offered earlier in life. Additionally, having a better understanding of the impact of iGBS disease on patients and families can help inform needed resources and services.

OBJECTIVES The purpose of the COMPPASS Registry is to establish a comprehensive data repository of patient, patient family, and provider reported outcomes and experiences, that will enhance research on the burden and impact of invasive Group B Streptococcus (iGBS), ultimately informing the development of evidence-based interventions and improving outcomes for at-risk and affected individuals and families.

SPECIFIC AIMS

Specific aims of the registry are to:

* Create a cohort of well-characterized patients with perinatal iGBS for participating in retrospective and prospective research
* Collect clinical and non-clinical data to support research to understand the range of neurodevelopmental impairment (NDI) associated with iGBS
* Collect clinical and non-clinical data to support research to understand the impact of iGBS disease on families of children affected by perinatal iGBS
* Collect parent and caregiver-reported patient outcomes following iGBS disease to improve care pathways and support services for affected individuals
* Improve awareness of and facilitate enrollment into clinical trials and research studies around perinatal iGBS and NDI

RESEARCH DESIGN AND METHODS The Registry will collect data globally on at least 10,000 children affected by perinatal iGBS over 10 years. It will gather information on the birthing parent's obstetric and pregnancy history, acute illness, postnatal discharge, neurodevelopmental outcomes, and family impact. Participants will consent to share de-identified information relating to these topics and complete validated surveys assessing neurodevelopmental impact at predetermined intervals. To be included in the registry, patients must be ill or had become ill from a group B strep infection at birth through the first 90 days of life and be between the ages of 0 and 19 years of age. In the instance of a multi-gestational pregnancy where at least one child has been diagnosed as having become ill from a Group B Strep infection, the similarly affected and/or unaffected sibling(s) will be invited to take part in the registry. Parents of children who were stillborn due to iGBS infection will also be invited to participate in the registry.

ENROLLMENT Parents or caregivers interested in taking part in the registry will be asked to complete a screening questionnaire to confirm they meet the inclusion criteria for the study. No identifiable information will be disclosed as part of the screening process.

Following the screener, the prospective participant will be asked to confirm their consent to take part in the study. Once the parent or caregiver's electronic consent has been obtained, a unique identifier will be automatically assigned to them and the iGBS-affected child (index child) by the system. Parents and caregivers will have the opportunity to provide information on siblings from multi-gestation pregnancies where at least one has been infected by iGBS infection and/or other sibling(s) affected by iGBS from other singleton pregnancies of same parent. A unique identifier will automatically be created for siblings which will be linked to the parent or caregiver, and the index child.

COLLECTION OF SUBJECT INFORMATION The Registry consists of a set of questionnaires and validated surveys to be completed by the parent or caregiver of the primary child and their sibling(s), where applicable. The list below outlines the questionnaires and surveys to be offered to participants for completion following consent.

Questionnaires The following retrospective questionnaires will be completed at baseline by either the parent or caregiver of the iGBS-affected child.

* Baby /Child Intake
* Demographics
* Obstetric History
* Pregnancy
* Postnatal Discharge

Surveys After completing the baseline questionnaires, parents and caregivers will be invited to participate in ongoing validated surveys. These optional surveys will be available at specific time points throughout the child's development, up to 18 years of age, with 1 to 5 surveys accessible at each time point.

To support discussions with healthcare providers, participants will also have the option to download their time-stamped responses upon completing each survey, providing valuable insights into their child's development over time.

The general frequency of surveys is as follows unless predefined by the survey owner:

Participant Age: 0-3 years | Survey Frequency: Every 3 months Participant Age: 4-5 Years | Survey Frequency: Every 6 months Participant Age: 6-18 Year | Survey Frequency: Once a year

The following validated neurodevelopmental surveys will be made available to registry participants:

* Ages & Stages Questionnaires®, Third Edition
* Ages & Stages Questionnaires®: Social-Emotional, Second Edition (ASQ®:SE-2)
* Child Behavior Checklist for Ages 11/2-5 Years
* Child Behavior Checklist for Ages for 6-18 Years
* Global Score for Early Development
* The Washington Group / UNICEF Child Functioning Module (CFM)
* The Washington Group / UNICEF Child Functioning Module (CFM)
* Higher Vision Function Question Inventory - Q11
* MacArthur-Bates Words and Gestures
* MacArthur-Bates Words and Sentences
* MacArthur-Bates CDI-III
* KIDSCREEN -27
* Beach Center Family Quality of Life Scale

FOLLOW-UP Participants will receive an email and/or text reminder of upcoming survey(s) a week before the survey availability window opens. The study team will have access to a completion status report of surveys which will support any additional engagement with participants who do not complete follow-up surveys.

PARTICIPANT RISK This Registry is an observational study; participants will not experience specific risks by participating. Participants may experience anxiety or psychological discomfort while completing the questionnaires and/or surveys. In addition, it is not possible to exclude with 100% certainty a breach of confidentiality by unauthorized parties gaining access to information included in electronic records. However, all reasonable safeguards to prevent loss of confidentiality have been undertaken. For instance, identifiable information will be stored separately from all other information gathered.

POTENTIAL BENEFITS Participants will receive no immediate benefit from participation in this study. Participants will be given access to their survey responses, which may be of benefit when discussing their child's development with healthcare professionals. Additionally, participation in this Registry may help increase understanding of how iGBS affects children and their families, leading to more research and awareness of families affected by prenatal iGBS.

ALTERNATIVES TO PARTICIPATION The alternative to participation in this study is not to participate in the Registry. If there are questions that the participant doesn't know the answer to, they have the option to select "I don't know".

WITHDRAWAL FROM PARTICIPATION Participants may withdraw from taking part in the Registry at any point in time and for any reason.

Participants may be withdrawn from the study for the following reasons:

1. Failure to complete the required study surveys, regardless of reason.
2. The child dies.

COSTS AND PAYMENTS All costs associated with the implementation and maintenance of the Registry shall be supported by Precia Group. Registry participants will incur no costs. Participants will not be compensated for their effort related to the Registry.

STATISTICAL CONSIDERATIONS AND REGISTRY REPORTING Because the Registry is not hypothesis-driven, formal prospective calculations of sample sizes are not provided. Instead, descriptive analyses will be conducted. We will periodically assess variation in iGBS-related NDI management, clinical events, and patient-reported outcomes to evaluate temporal changes concurrent with registry participation.

Assessments will be made on general population characteristics, frequency of missing data, and elements to support quality control of the data being entered into the Registry.

ELIGIBILITY:
Inclusion Criteria:

1. A child below the age of 19 who was either diagnosed with or received a lab test result confirming an iGBS infection, or being able to describe their child's condition and experience with iGBS infection at, or within 90 days of, birth.

   or A child who was diagnosed as having invasive Group B Strep infection within the first 90 days after delivery and later passed away because of the infection or Parent who has experienced a stillbirth due to iGBS infection
2. A sibling(s) from a multi-gestation pregnancy where at least one child was diagnosed as having invasive Group B Strep infection
3. Parent or caregiver who understands and electronically signs the inform consent document
4. In addition to parental or caregiver consent, children between the ages of 13-17 years who are able to understand and provide assent to take part in the study, as confirmed by an electronic signature by their consenting parent or caregiver.

Exclusion Criteria:

1. A child affected by iGBS infection currently over the age of 18.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child(ren) who are ill or had become ill from a Group B Streptococcus infection at birth through the first 90 days of life and be between the ages of 0 and 19 years of age. In the instance of a multi-gestational pregnancy where at least one child has been diagnosed as having become ill from a Group B Strep infection, the similarly affected and/or unaffected sibling(s) will be invited to take part in the registry. Information from parents of children who were stillborn will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2035-03-31 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Stillbirth Due to Invasive Group B Streptococcus | After 20 weeks gestation to the delivery of fetus
  Intrauterine fetal death
Parent or Care-giver Reported Diagnosis of Early-Onset Invasive Group B Streptococcus | Within 24 Hours of Birth
Parent or Caregiver Reported Diagnosis of Late-Onset Invasive Group B Streptococcus | Up to 90 Days after Birth

CONTACTS AND LOCATIONS:
Overall Officials: Donna Russell, MPA, Principal Investigator — Precia Group

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with approved investigators.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication date
Access Criteria: Access to de-identified registry data may be granted upon request to the Scientific Advisory Board and the Registry Data Access Committee.